CLINICAL TRIAL: NCT02569372
Title: A Prospective, Open-label, Dose-escalation, Single-center, Phase I Trial to Explore the Tolerability, Safety and Pharmacokinetics/Pharmacodynamics of GC1102 (Recombinant Hepatitis B Human Immunoglobulin)
Brief Title: A Phase 1 Study of GC1102 (Recombinant Hepatitis B Immunoglobulin) in Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC1102B_P1
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- GC1102 80,000 IU(Single does) (Experimental): GC1102 80,000 IU(Single does) I.V.
  Interventions: Biological: GC1102
- GC1102 120,000 IU(Single does) (Experimental): GC1102 120,000 IU(Single does) I.V.
  Interventions: Biological: GC1102
- GC1102 180,000 IU(Single does) (Experimental): GC1102 180,000 IU(Single does) I.V.
  Interventions: Biological: GC1102
- GC1102 240,000 IU(Single does) (Experimental): GC1102 240,000 IU(Single does) I.V.
  Interventions: Biological: GC1102
- GC1102 80,000 IU(Multiple does) (Experimental): GC1102 80,000 IU(Multiple does) I.V.
  Interventions: Biological: GC1102
- GC1102 120,000 IU(Multiple does) (Experimental): GC1102 120,000 IU(Multiple does) I.V.
  Interventions: Biological: GC1102
- GC1102 180,000 IU(Multiple does) (Experimental): GC1102 180,000 IU(Multiple does) I.V.
  Interventions: Biological: GC1102
- GC1102 240,000 IU(Multiple does) (Experimental): GC1102 240,000 IU(Multiple does) I.V.
  Interventions: Biological: GC1102

INTERVENTIONS:
Biological: GC1102 — GC1102(Recombinant Hepatitis B Human Immunoglobulin)

SUMMARY:
This study is SAD(Single Ascending Dose)/MAD(Multiple Ascending Dose) study to Explore the Tolerability, Safety and Pharmacokinetics/Pharmacodynamics of GC1102 (Recombinant Hepatitis B Human Immunoglobulin) in Chronic Hepatitis B Patients.

DETAILED DESCRIPTION:
GC1102 is a new recombinant hepatitis B human immunoglobulin. This study is composed with 2 Parts, Part A for SAD and Part B for MAD and total 4 dosing program which is escalated after confirming safety. Maximum 48 subjects will be participated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis B or those who diagnosed with chronic hepatitis B carrier who given written informed consent.
* Patients aged ≥19 and ≤ 65 years
* If Naïve for the Nucleos(t)ide analogs therapy, HBeAg (-), HBsAg 1,000 IU/mL or less and HBV DNA 2,000IU/mL or less Or If currently receiving Nucleos(t)ide analogs therapy, HBeAg (±), HBsAg 1,000 IU/mL or less and HBV DNA (-: limit of detection of 60 IU/mL or less).

Exclusion Criteria:

* Patients who currently involved or has participated in any other clinical trial within 30 days.
* Patients co-infected with HAV, HCV or HIV
* Patients with history of malignant tumor within 5 years except basal cell carcinoma of skin, cervical intraepithelial neoplasia.
* Patients who have active infection except chronic hepatitis infection.
* Patients with liver disease who had complications such as gastroesophageal variceal, ascites and hepatic encephalopathy.
* Having eGFR 59 mL/min/1.73m2 or less with MDRD Evaluation phase (moderate reduction in GFR or more )
* Having blood or protein 1+ or more by the urine analysis with microscopic examination.
* Patients who have a clinically significant kidney disease including glomerulonephritis, anuria, acute renal failure, dialysis and renal transplantation.
* Patients with Vasculitis.
* Having leukocytes <3.0 x109/L
* Having Absolute Neutrophil Count<1.5x109/L
* Having platelet <750,000/mm3 during screening
* Having hemoglobin <10g/dL
* Having positive sign of serum cryoglobulin level.
* Having serum anti-nuclear antibody (ANA) 1:160 or more
* Patients who showed positive sign of serum perinuclear anti-Neutrophil Cytoplasmic Antibodies (p-ANCA).
* Patients who showed positive sign of serum cytoplasmic anti-Neutrophil Cytoplasmic Antibodies (c-ANCA).
* Patients who had history or be suspected of immune disease
* Patients who had experienced cardiovascular attack, myocardiac infarction, heart failure, PTCA or coronary artery bypass, angina, arrhythmia, any other clinically meaningful valvular heart disease, cerebral infarction or cerebral hemorrhage within 6 months.
* Patients who had history of anaphylaxis against the main component or subcomponent of study drug.
* Patients who had been administered live vaccine parentally (measles vaccine, parotitis vaccine, rubella vaccine, cholera combined vaccine, varicella vaccine) within 3 months prior to the dosing of study drug.
* Patients who had been received an immunosuppressant, immunity-modifying drug including interferon agents, cytotoxic chemotherapy that can affect their immune system, or radiation therapy within 3 months prior to the dosing of study drug
* Patients who had been treated with any other immunoglobulin within 3 months prior to the dosing of study drug
* Patients who had been treated with systemic steroid Therapy(more than 20 mg/day of prednisolone or its equivalence administered every day for more than 14 days, or more than 700 mg of a cumulative dose during the same period of time) within 3 months prior to the dosing of study drug (topical administration such as topical ointments, eye drops, inhalants or intranasal use, intra-articular injection, or tendon injection is acceptable; alternative-day treatment is acceptable even though administered for more than 14 days)
* Women who showed positive sign of pregnancy test before administered study drug.
* Those who do not agree to use appropriate contraceptive methods (condom, diaphoretic, an intrauterine device, oral contraceptive hormones, or a vasectomy of male sex partner) during the clinical trials.
* Those who had experienced bleeding more 400ml or a blood donation within 8 weeks prior to the dosing of study drug.
* Those who had been abused alcohol or any other drug within 6 months.
* Those who are judged disqualified to join clinical trials by investigator for other clinically significant medical or psychiatric condition.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity after the administration of GC1102 | Part A: 4weeks, Part B: 7 weeks
Adverse events after the administration of GC1102 | Part A: 4weeks, Part B: 7 weeks
Clinical findings in physical examination, vital signs and clinical laboratory after the administration of GC1102 | Part A: 4weeks, Part B: 7 weeks

SECONDARY OUTCOMES:
HBsAg sero-conversion rate from positive to negative after the administration of GC1102 till End of Study visit | Part A: 4weeks, Part B: 7 weeks
Geometric mean titer of serum HBsAg at each measurement point after the administration of GC1102 | Part A: 4weeks, Part B: 7 weeks
Geometric mean titer of serum HBV DNA of each measurement point after the administration of GC1102 | Part A: 4weeks, Part B: 7 weeks
Occurrence rate of anti-GC1102 antibody | Part A: 4weeks, Part B: 7 weeks
Occurrence rate of HBV DNA sequence changes after the administration of GC1102 | Part A: 4weeks, Part B: 7 weeks

OTHER OUTCOMES:
Ctrough for Part B | 7 weeks
Terminal elimination half-life (t½β) | Part A: 4weeks, Part B: 7 weeks
Area under the time concentration curve from 0 to last and infinity (AUClast, AUC0-∞) | Part A: 4weeks, Part B: 7 weeks
Maximum plasma concentration(Cmax) | Part A: 4weeks, Part B: 7 weeks
Time to maximum plasma concentration (Tmax) | Part A: 4weeks, Part B: 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hoon An, M.D., Principal Investigator — Severance Hospital; Chin Kim, Study Director — Green Cross Corporation
Locations (1):
- Severance Hospital, Seoul, South Korea